CLINICAL TRIAL: NCT01314573
Title: The Impact of High Intensity Exercise Upon EPC Number and Function in Young Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Dr. Karen Birch, University of Leeds, Sport and Exercise Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOSCI-10-007
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Exercise Anaphylaxis
Keywords: High intensity exercise training; Vascular health; Endothelial function; Circulating angiogenic cells; endothelial progenitor cells; Aerobic capacity; Arterial stiffness; Traditional and emerging cardiovascular disease risk factors
MeSH Terms: conditions — Exercise-Induced Allergies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interval maximal exercise (Experimental): Interval exercise involving repeated Wingate tests (30s durations of maximal exercise on a cycle ergometer).
  Interventions: Behavioral: Sprint interval exercise
- Continuous maximal exercise (Experimental): Continuous exercise of maximal exertion that has been work matched to an initial bout of interval exercise of 4 x 30s of maximal exercise. This exercise is performed on a cycle ergometer.
  Interventions: Behavioral: Maximal continuous exercise

INTERVENTIONS:
Behavioral: Sprint interval exercise — 3 session per week of exercise on a exercise cycle ergometer. Each session involves 30s of maximal exercise followed by 4.5 min of easy cycling at 10W. This is repeated 4 times at each exercise session.
  Other Names: high intensity exercise training
  Arms: Interval maximal exercise
Behavioral: Maximal continuous exercise — 3 sessions per week of an exercise intervention involving maximal cycling until the participant has completed an amount of work equivalent to a sprint interval training session. This exercise lasts between 3 and 3.5 minutes.
  Other Names: high intensity exercise training
  Arms: Continuous maximal exercise

SUMMARY:
The purpose of the study is to examine the effects of different exercise intensity training programs upon blood vessel function and circulating blood cells involved in blood vessel repair in young women. The long term effects of exercise may be beneficial to cardiovascular health and it is important to understand the training methods that are the most beneficial. In particular we aim to determine if brief maximal exercise improves the function and stiffness of blood vessels and enhance blood vessel repair. Two methods of exercising are being compared, exercise bouts involving intermittent exercise and exercise completed all at once, but at a very high intensity.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy females
* Between 18-25 years old
* No on medication (this includes contraceptives)

Exclusion Criteria:

* Medication use (including oral contraceptives)
* Amenorrhoea
* High blood pressure
* Very active (>3 hours per week of organized physical activity)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake | 4 weeks
  A measure of aerobic capacity determined during an incremental exercise test to volitional fatigue on an exercise ergometer.

SECONDARY OUTCOMES:
Heart rate variability | 4 weeks
Endothelial progenitor cell function | 4 weeks
  measures of in vitro cell migratory ability, adhesion and classification of endothelial progenitor cells
Flow mediated dialtion | 4 weeks
  Measure of vascular endothelial function determined non-invasively at the brachial artery
Arterial stiffness | 4 weeks
  The stiffness of the carotid artery is measured using a combination of ultrasound imaging and non-invasive blood pressure measurements. Lower degrees of stiffness are more favourable.
Circulating angiogenic cell numbers | 4 weeks
  These cells are involved in vascular repair and proliferation and may be measured using flow cytometric methods. Specifically cells with CD34 and CD309 antigens are enumerated.
Endothelial progenitor cell function | 4 weeks
  Measure of in vitro migratory, adhesion and classification of endothelial progenitor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Birch, BSc PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom